CLINICAL TRIAL: NCT06059755
Title: Comparison of Mirror Therapy Versus Cross- Education Non Paretic Limb Training on Upper Limb Strength and Hand Dexterity in Stroke Survivors.
Brief Title: Mirror Therapy vs Cross Education Non Paretic Limb Training on Strength and Hand Dexterity in Stroke Survivors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Kainat Rashid
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hemiplegia and Hemiparesis
Keywords: Paresis, Mirror therapy, Motor skills, Stroke
MeSH Terms: conditions — Hemiplegia; Paresis; Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Cross education (Experimental): For strength training resistance exercises with a load of 60% of one repetition maximum will be performed targeting the muscles involved in upper limb function. It includes exercises like shoulder presses, wrist curls, elbow flexion, and triceps extensions. Among the functional movements that are the focus of motor skill training activities for non-paretic limbs are reaching, gripping, and object manipulation. Patient will be encouraged to mentally visualize themselves performing movements and tasks with the affected limb, while actively engaging the non-paretic limb. Strength will be measured using the grip strength test/ hand held dynamometer. Patients will undergo 45-minute session per day, 3 days per week for 6 weeks.
  Interventions: Other: Cross education
- Group B: Mirror Therapy (Experimental): Participants will be asked to sit in front of a table of appropriate height with their arms resting on the table and a mirror (35 cm × 35 cm) placed between the patient's arms. The non-affected arm will be placed in front of the mirror and the affected arm will be placed and obscured. Patient will engage in specific exercises or movements using the affected limb while observing the mirror reflection. The movements will consist of forearm rotation, elbow, wrist, and finger flexion and extension movements, and hand grasping. Appropriate movement tasks will be selected according to the function of the affected upper limb. This exercise will be performed 45 minutes per day, 3 times per week for 6 weeks.
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Cross education — For strength training resistance exercises with a load of 60% of one repetition maximum will be performed targeting the muscle involved in upper limb function. Strength will be measured using the grip strength test/hand held dynamometer. Patients will undergo 45 minute session per day, 3 days per week for 6 weeks.
  Arms: Group A: Cross education
Other: Mirror Therapy — Participants will be asked to sit in front of a table of appropriate height with their arms resting on the table and a mirror (35 cm × 35 cm) placed between the patient's arms. The non-affected arm will be placed in front of the mirror and the affected arm will be placed and obscured. Appropriate movement tasks will be selected according to the function of the affected upper limb. This exercise will be performed 45 minutes per day, 3 times per week for 6 weeks
  Arms: Group B: Mirror Therapy

SUMMARY:
A stroke is a significant contributor to functional decline and long-term disability. The reduction of obesity and improvement in quality of life are directly correlated. Many post-stroke patients experience persistent upper extremity dysfunction. The study aims to compare cross-education non-paretic limb training versus mirror therapy on upper limb strength and dexterous movement of hand in stroke survivors This randomized clinical trial will be conducted at DHQ Hospital Sargodha over a duration of six months. The sample size will consist of 26 participants. Participants which meet the inclusion criteria will be selected through Non probability convenience sampling technique, which will further be randomized through computer engendered in blocks by using basic number generator.13 participants will be assigned to Cross education group and 13 participants will be assigned to Mirror Therapy group. Data will be using various assessment tools, including the Action Research Arm Test (ARAT) for functional limitation, Fugl-Meyer Assessment-upper extremity (FMA-UE), Stroke Impact Scale (SIS) for hand dexterity and function. Hand held dynamometer will be used for Grip Strength Test. Pre intervention assessment will be conducted for both groups. The effects of intervention will be measured at pretreatment ,3rd week and post intervention. Data analysis will be performed by using SPSS (Statistical Package for Social Sciences) 23 version.

DETAILED DESCRIPTION:
A stroke or CVA is characterized by the sudden onset of focal neurological dysfunction symptoms that persist for more than 24 hours (or cause death earlier) and are brought on by an acute vascular injury to a specific area of the brain. Overall, a stroke creates a blockage in the delivery of blood and oxygen to a particular region of the brain, which results in cell death, long-term or lifelong impairments, or even death. Issues with paralysis, motor control, pain-related sensory problems, language usage or comprehension, thinking, memory, and emotional challenges are just a few examples of disabilities.

Stroke can be ischemic or hemorrhagic. Over 100 diseases are associated with ischemic stroke, making it heterogeneous. It is the most common type of stroke and accounts for 87% of all strokes. Ischemic stroke is further divided into two groups; thrombotic stroke (the formation of clot or plaque in blood vessels within the brain) and embolic stroke (the formation of clot or plaque somewhere else in the body and travels to blood vessel of the brain through blood stream).

Atherosclerosis, arterial dissection, and artery-to-artery embolism are all examples of large vessel disease. The primary small vessel diseases causing lacunar strokes are lipohyalinosis and atherosclerosis. Intracerebral hemorrhage, which can occur deep (basal ganglia, brainstem), cerebellum, or lobar, accounts for about 15% of strokes. About 20% of intracerebral hemorrhages are brought on by macro vascular lesions (vascular malformations, aneurysms, cavernomas), venous sinus thrombosis, or other uncommon causes; these are particularly significant in young patients.

Literature review A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines. Search term for the initial literature review was post-stroke mirror therapy, post-stroke cross education, comparison of mirror therapy versus cross education non paretic limb training, upper limb strength and hand dexterity.

O. van der Groen et al. (2023) studied the Corticospinal and intracortical responses from both motor cortices following unilateral concentric versus eccentric contractions and compared responses to transcranial magnetic stimulation(TMS) in both motor cortices following single sessions of unilateral ECC and CON exercise of the elbow flexor and concluded that These findings suggest that responses after a single bout of exercise may not reflect longer term adaptations.

S. Karamat et al. (2022) compared the effects of task-based mirror therapy and Repetitive Facilitation Exercise on upper limb function in post stroke patient. The study concluded that mirror therapy and repetitive facilitation Exercise both were found to be effective in improving upper limb motor functions of acute stroke patients. However, Mirror therapy has shown significant effects in upper extremity functional index.

ELIGIBILITY:
Inclusion Criteria:

* • Age range between 45-65 years.

  * Both male and female genders.
  * Clinically diagnosed of stroke referred by Neuro physician.
  * Patients in the subacute stage, duration of 3 to 6 months from onset.
  * Patients with anterior cerebral artery (ACA) and middle cerebral artery (MCA) involvement with the affected side being the dominant side.
  * Patients with Mini-Mental State Examination (MMSE) score more than 16.
  * According to Modified Ashworth Scale, patients in range of 1 and 1+ (Flexor carpal radialis muscle,Flexor carpal ulnaris muscle, Flexor digitorum profundus muscle, Flexor digitorum superficialis muscle, Flexor pollicis longus muscle, Palmaris longus muscle) will be included .
  * Hemiparesis or hemiplegic due to Ischemic stroke

Exclusion Criteria:

* Patients with Alzheimer disease, Parkinson's disease, Multiple sclerosis and Brain tumors .
* Those with severe cognitive impairment , those who were unable to provide informed consent. Patients having acute pericarditis, lumbar puncture within 7 days, Major surgery or major trauma within 14 days.
* Patient with recurrent stroke.
* With unilateral neglect or apraxia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (For Functional Limitation) | Changes from baseline Action Research Arm Test at 3rd week and after 6 weeks
  The instrument contains 19 items grouped into 4 subtests; grasp, grip, pinch, and gross motor. Item performance is rated on a 4-point scale (0=unable; 1=partial; 2= abnormal; 3=normal) then item ratings are summed and reported out of 57 points with higher score indicating greater UE function.
Fugl-Meyer Assessment. (For Upper extremity function) | Changes from baseline Fugl-Meyer Assessment at 3rd week and after 6 weeks
  The Fugl-Meyer Assessment is the gold standard to assess motor function of post-stroke hemiparesis. The FMA-UE consists of 30 items assessing motor function and 3 items assessing reflex function. The scores most applicable to task performance is given from "0, inability," "1, beginning ability," to "2, normal" (total score range, 0-66).Higher the score more is the independence.
Hand-held dynamometer. (For Upper Limb strength assessment) | Changes from baseline Fugl-Meyer Assessment at 3rd week and after 6 weeks
  This instrument is scored using force produced in kilograms (0-90) or pounds (0-200). The subject is seated with back, pelvis and knees as close to 90 degrees as possible, shoulder is adducted and neutrally rotated, elbow flexed to 90 degrees, and forearm neutral and wrist held between 0-15 degrees of ulnar deviation. Maximum grip is the mean of 3 trails.
Stroke Impact Scale (For hand function) | Changes from baseline Fugl-Meyer Assessment at 3rd week and after 6 weeks
  The Stroke Impact Scale (SIS) is a stroke-specific, self-report, health status measure. It contains 59 items and assesses 8 domains: Strength - 4 items, Hand function - 5 items, ADL/IADL - 10 items, Mobility - 9 items, Communication - 7 items, Emotion - 9 items, Memory and thinking - 7 items, Participation/Role function - 8 items. For each item individual is asked to rate the level of difficulty in past two weeks using the scale;1= extremely difficult, 2= very difficult, 3= somewhat difficult, 4= a little difficult, 5= not difficult at all. On a scale of 0 to 100, with 100 representing full recovery and 0 representing no recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Kianat Rashid, MSPT-NM, Principal Investigator — Riphah International University
Locations (1):
- Tehreem Mukhtar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No